CLINICAL TRIAL: NCT04347356
Title: Relationship of Balance, Functional Capacity, Fear of Movement and Quality of Life With Lower Extremity Muscle Strength in Elderly People
Brief Title: Relationship of Balance, Functional Capacity and Fear of Movement With Lower Extremity Muscle Strength in Elderly
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BVUsozyilmaz01
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Elderly
Keywords: Balance; elderly; fear of movement; functional capacity; lower extremity muscle strength; quality of life
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aging is a period in which the morphological, physiological and pathological changes progress negatively, accompanied by various diseases and regression of physical and mental abilities. In this period, the individual experiences biological and physiological losses as well as social problems in his/her life. From the age of 65, approximately 80% decrease in muscle strength can be observed and this decrease is especially noticeable in the leg and trunk muscles. Decreases in the strength of the muscles in the lower extremities may cause deterioration in physical function, decrease in mobility, increase in falling related accidents, also can cause osteoporosis and physical deficiencies. Determining the structures with which the lower extremity muscle strength is related will facilitate the precautionary measures for the inadequacies that will arise in the later stages of aging.

This study was performed to analyze the relationship of lower extremity muscle strength with balance, functional capacity, fear of movement and quality of life in elderly individuals living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be 65-88 years old,
* The participant must have a minimus score of 24 on the Mini-Mental State Examination (MMSE),
* No cognitive impairment,
* The participant must be independent of daily life activities (must not use an assistive device for walking).

Exclusion Criteria:

* Having a disease that can affect balance (vestibular, neurological, orthopedic ...) performing regular exercise
* Uncontrolled hypertension or arrhythmia
* Uncontrolled diabetes mellitus
* Orthopedic, neurological or musculoskeletal problems
* Postural hypotension
* Obesity (body mass index>40)
* Uncompensated clinical conditions such as chronic obstructive pulmonary disease, interstitial lung disease, heart failure, or rheumatic and psychiatric diseases

Ages: 65 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects aged between 65-88 years who are a minimum score of 24 on the Mini-Mental State Examination, no cognitive impairment, and are independent of daily life activities will be included in the study.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Muscle Strength | Baseline
  Lower limb muscle strength will be assessed by sit-to-stand test. Participants will be asked to perform sit-to-stand maneuver as fast as possible for 30 seconds and the number of completed repetitions will be recorded.
Static Balance | Baseline
  Static balance will be assessed by single leg stance test. The time that patients can remain in balance on the dominant leg with their eyes open is recorded. Time under 10 seconds indicates loss balance.
Dynamic Balance | Baseline
  Dynamic balance will be assessed by the Timed Up and Go Test. The TUG measures the time it takes for a participant to stand up from a standard chair, walk 3m, turn, walk back to the chair, and sit down again. The cut-off score of 12 seconds in older persons is the threshold value for an increased risk of falling.
Postural Balance | Baseline
  The postural balance will be assessed by the Berg Balance Scale. It assesses 14 functions related to daily activities. A score of 0 represents an inability and a score of 4 represents independently. The maximum score is 56. A score of less than 45 indicates balance loss.
Fear of Movement | Baseline
  Fear of movement will be assessed by the Tampa Scale for Kinesiophobia. Individuals get a minimum of 17 and a maximum of 68 points. A high score indicates an increasing degree of kinesiophobia.

SECONDARY OUTCOMES:
Functional Capacity | Baseline
  Functional capacity will measured with the 6-minute walk test.Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society (ATS).
Notthingham Health Profile Assesment | Baseline
  The quality of life will be assessed by Notthingham Health Profile. The minimum score is '0', the maximum score is '100'. "0 score" shows the best health, "100 score" shows the worst health.

CONTACTS AND LOCATIONS:
Overall Officials: Semiramis Ozyilmaz, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)